CLINICAL TRIAL: NCT00452101
Title: Randomized, Placebo Controlled Trial: Effects of Aquamin F Alone or in Combination With Glucosamine Sulfate on Joint Mobility and Pain in Osteoarthritis of the Knee
Brief Title: Effects of Aquamin F on Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Marigot Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MARC005-065
Record Dates: First submitted 2007-03-22; First posted 2007-03-26 (Estimated); Last update posted 2007-03-26 (Estimated); Status verified 2007-03

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Clinical trial; Aquamin F; Glucosamine
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aquamin F

SUMMARY:
The objective of this trial is to evaluate the effect of Aquamin F alone or in combination with glucosamine sulfate versus placebo on symptoms of joint pain, stiffness and immobility in subjects with painful osteoarthritis of the knee. The following hypotheses were tested:

(Hypothesis 1) After 12 weeks of treatment, subjects taking Aquamin F alone or in combination with glucosamine sulfate will have significantly less joint pain, stiffness and immobility compared to subjects taking glucosamine sulfate alone or placebo alone.

(Hypothesis 2) No significant differences will be seen for adverse events between the subjects taking Aquamin F, glucosamine sulfate, Aquamin F + glucosamine sulfate or placebo.

DETAILED DESCRIPTION:
Method: Subjects were randomized to receive 12 weeks of Glucosamine sulfate vs Aquamin F vs Placebo vs Aquamin F + Glucosamine sulfate while controlling for pain with acetaminophen. Subjects were then followed for blood chemistry measurements only over an additional 12-week period specifically to assess blood calcium levels post treatment. All participants were subjected to the same diet and exercise regimen and measurements included: WOMAC scores (pain, stiffness, mobility, total score), 6 Minute Walking Distances, active and passive range of motion measurements, DXA scans, blood chemistry, hematology, CRP levels and lipid profiles as well as rescue medication diary measurements and adverse event assessments. An independent statistician analyzed the data using independent t-tests and ANCOVA for between-group comparisons and matched-pair t-tests for within-group comparisons of patients included in ITT-LOCF and completer analyses.

ELIGIBILITY:
Inclusion Criteria

* Subjects aged 35 to 75, male or female
* Subjects diagnosed with symptomatic moderate to severe osteoarthritis of the knee according to the modified criteria of the American College of Rheumatology17, 18
* Subjects who present with osteoarthritis of the knee as judged by symptoms and disabilities detectable through published, validated questionnaires or previous diagnosis by a physician.
* Subjects who are symptomatic with daily or near daily pain and stiffness from osteoarthritis.
* Subjects with screening WOMAC Osteoarthritis Index total score (transformed score) of not more than 75.
* Subjects with ability to comprehend and complete the questionnaires and forms.
* Subjects whose schedules permit clinic evaluations every four weeks.
* Subjects who are willing to stop taking calcium supplements, if any, and to restrict consumption of high calcium foods to 600 mg (two dairy serving) per day
* Subjects with a high probability of compliance with study procedures and test article consumption.
* Subjects willing and able to follow protocol guidelines and schedules, and complete diaries.
* Subjects who are likely to abstain from taking unauthorized supplements or participating in any other clinical trial or experimental treatment during this trial
* Subjects with normal gastrointestinal digestion and absorption.

Exclusion Criteria

* Subjects suffering from inflammatory arthritis, gout, pseudogout, Paget's disease, seizure disorder, insulin dependent diabetes mellitus, uncontrolled hypertension, unstable cardiovascular disease, active hepatic or renal disease, active cancer and/or HIV infection.
* Subjects who are non-ambulatory or bedridden due to osteoarthritis.
* Subjects who are dependent on prescription drugs to control pain.
* Subjects on any other clinical trial or experimental treatment in the past 3 months
* Subjects who are pregnant, lactating, or at risk of becoming pregnant.
* Subjects who have received:

  * Non-Steroidal Anti-Inflammatory Drugs (NSAIDS) within 48 hours prior to study enrollment.
  * Intramuscular or systemic corticosteroid injection within 4 weeks prior to study enrollment.
  * Intra-articular corticosteroid injection within 2 months prior to study enrollment.
  * Intra-articular hyaluronic acid injection within 4 months prior to study enrollment.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2006-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
WOMAC scores (pain, stiffness, mobility, total score)
6 Minute Walking Distances
Active and passive range of motion (goniometer measurements)

SECONDARY OUTCOMES:
DXA scans for bone mineral density
CRP levels
Lipid profiles
Rescue medication diary measurements
The safety/toxicology measurements included a Chemistry Profile (including serum calcium)
Complete Blood Counts
Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: John L Zenk, MD, Study Chair

REFERENCES:
- [Derived] Frestedt JL, Walsh M, Kuskowski MA, Zenk JL. A natural mineral supplement provides relief from knee osteoarthritis symptoms: a randomized controlled pilot trial. Nutr J. 2008 Feb 17;7:9. doi: 10.1186/1475-2891-7-9. PMID 18279523